CLINICAL TRIAL: NCT03313297
Title: A Double-blind, Randomized, Placebo-controlled Phase II Pilot Trial Investigating Efficacy, Safety and Feasibility of 11β-hydroxysteroid Dehydrogenase Type 1 Inhibition by AZD4017 to Improve Skin Function and Wound Healing in Patients With Type 2 Diabetes
Brief Title: Glucocorticoids and Skin Healing in Diabetes (GC-SHealD)
Acronym: GC-SHealD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Ana Tiganescu, PhD, Scientific Lead, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ED17/93260
Record Dates: First submitted 2017-10-05; First posted 2017-10-18 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: skin; wound healing; 11 beta-hydroxysteroid dehydrogenase type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 2-(1-(5-(cyclohexylcarbamoyl)-6-propylsulfanylpyridin-2-yl)-3-piperidyl)acetic acid

STUDY DESIGN:
Intervention Model Description: Double-blind, randomised, parallel group, placebo-controlled phase II pilot trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment groups will be allocated in a double-blind manner. Participants will be blinded to the treatment they receive (placebo or drug) throughout all stages of the study. Investigators will also be blinded to the treatment until all samples have been collected and processed. Blinding will be generated by a dedicated trials pharmacy representative who is not otherwise associated with this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZD4017 (Active Comparator): 400mg oral AZD4017 twice daily for 35 days
  Interventions: Drug: AZD4017
- Placebo (Placebo Comparator): A placebo tablet containing microcrystalline cellulose and sodium stearyl fumarate to match the active tablets in size, shape and colour.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD4017 — AZD4017 is a novel orally bioavailable small molecule inhibitor of 11β-HSD1 enzyme activity. It is potent and highly selective in vitro and in vivo. The half maximal inhibitory concentration (IC50) for inhibition of 11β-HSD1 activity (cortisone to cortisol conversion) is 2nM. AZD4017 is selective (> 2000x) for 11β-HSD1 over human recombinant 11β-HSD2 and the closely-homologous enzymes 17β-hydroxysteroid dehydrogenase 1 and 17β-hydroxysteroid dehydrogenase 3 in vitro.
  Arms: AZD4017
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
The study aims to investigate effects of inhibiting glucocorticoid activation on skin function and wound healing in patients with type 2 diabetes. Half of patients will be given a drug to inhibit glucocorticoid activation and the other half will be given a placebo.

DETAILED DESCRIPTION:
Glucocorticoids are known to impair skin function and wound healing which are also compromised in patients with type 2 diabetes. The enzyme 11 beta-hydroxysteroid dehydrogenase type 1 (11β-HSD1) activates glucocorticoids in target tissues including skin. Pre-clinical data demonstrate that 11β-HSD1 inhibition improves skin function and wound healing but this has not been investigated in man.

Using the 11β-HSD1 inhibitor AZD4017, we will investigate if

1. Oral AZD4017 inhibits 11β-HSD1 activity in skin
2. AZD4017 is safe and well-tolerated in patient with T2DM
3. Oral AZD4017 regulates skin function
4. Systemic glucocorticoid levels and skin 11β-HSD1 activity, independently or in combination correlate with measures of skin function

Study feasibility will also be assessed; if successful, data from this pilot study will inform power calculations for a future trial to investigate the ability of 11β-HSD1 inhibition to promote foot ulcer healing in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to consent
2. Type 2 diabetes with HbA1c ≤11% (≤97 mmol/mol) at screening while taking standard therapy at a stable dose for ≥10 weeks

Exclusion Criteria:

1. Women of child-bearing potential
2. Active leg/foot ulceration
3. Clinically relevant acute electrocardiogram anomalies
4. Uncontrolled hypertension
5. Endocrine disorder (other than type 2 diabetes ), including type 1 or secondary diabetes (except treated hypothyroidism)
6. Gilbert's disease
7. Alanine aminotransferase and/or aspartate aminotransferase and/or alkaline phosphatase >1.5x upper limit of normal (ULN)
8. Bilirubin >1.5x ULN
9. Estimated glomerular filtration rate <45 ml/min/m2
10. Creatine kinase >2x ULN
11. Drug abuse within the last year
12. Any glucocorticoid treatment within 3 months of screening
13. Anti-coagulant medication
14. Probenecid therapy
15. Medical/surgical procedure or trauma during drug administration or one week after drug cessation (excluding skin biopsies)
16. Involvement in trial planning and/or conduct
17. Participation in other clinical study within 1 month
18. Deemed inappropriate to participate by the trial team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Skin 11β-HSD1 activity | Change between day 0 and day 28
  Enzyme activity radioassay to evaluate AZD4107 efficacy in skin

SECONDARY OUTCOMES:
Urinary cortisol / cortisone metabolites | Change between day 0 and day 35
  Urine samples for tetrahydrocortisol / tetrahydrocortisone metabolite ratios to evaluate systemic AZD4107 efficacy
AZD4017 in plasma | Change between day 0 and day 28
  Quantification of AZD4017 concentration in plasma to evaluate systemic AZD4107 exposure
AZD4017 in skin | Change between day 0 and day 28
  Quantification of AZD4017 concentration in plasma to evaluate skin AZD4107 exposure
Discontinuation due to Adverse Event | Day 42
  Adverse Event-related participant withdrawals to evaluate safety
Body mass index | Change between day 0 and day 35
  Body mass index to evaluate safety
Waist-hip ratio | Change between day 0 and day 35
  Waist-hip ratio to evaluate safety
Blood pressure (sphygmomanometer) | Change between day 0 and day 35
  Blood pressure to evaluate safety
Sudomotor function | Change between day 0 and day 35
  Conducted with a Sudoscan device to measure c-fiber innervation in hands and feet for skin function
Skin hydration | Change between day 0 and day 35
  Conducted with a Corneometer device to measure skin water content for skin function
Epidermal barrier function | Change between day 0 and day 35
  Conducted with a Tewameter device to measure skin trans-epidermal water loss for skin function
Epidermal barrier integrity | Change between day 0 and day 28
  Conducted by tape tripping to a pre-determined trans-epidermal water loss rate for skin function
Skin thickness | Change between day 0 and day 35
  Conducted by Optical Coherence Tomography imaging for skin function
Wound healing | Change between day 0 and day 2
  Conducted by Optical Coherence Tomography imaging for skin function
Wound healing | Change between day 0 and day 7
  Conducted by Optical Coherence Tomography imaging for skin function
Wound healing | Change between day 28 and day 30
  Conducted by Optical Coherence Tomography imaging for skin function
Wound healing | Change between day 28 and day 35
  Conducted by Optical Coherence Tomography imaging for skin function
Skin RNA-seq gene expression profiling | Change between day 0 and day 28
  For skin function

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals Trust, Leeds, United Kingdom